CLINICAL TRIAL: NCT03350672
Title: Validation of a Urine Assay to Measure Tenofovir Levels in Patients Taking Tenofovir Alafenamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Philadelphia Fight (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PhiladelphiaFight
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hiv
Keywords: HIV prevention; PrEP; Descovy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: 1a) Ten healthy subjects will be given seven daily doses of TAF/FTC under direct observation to ensure adherence.
  1b) Ten healthy subjects will be given one daily dose of TAF/FTC under direct observation to ensure adherence. Morning (not first morning) urine and plasma samples will be collected starting the day the dose is given (1 hr post-dose) and every day thereafter for 6 days.
  2) Ten HIV-positive patients who have had undetectable viral loads for greater than 12 weeks (and a recent undetectable viral load in the previous 4 weeks) on an antiretroviral regimen containing TAF/FTC (i.e. Genvoya™, Odefsey™, or Descovy™ in combination with another HIV medication or medications) will have one-time pre-dose urine (early morning) and plasma samples drawn for tenofovir (TFV) concentration, as well as a comprehensive metabolic panel for measurement of creatinine clearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1a (Experimental): Age 18 or older at the time of signed informed consent
  * Not currently taking commercial FTC/TDF for PrEP or any other investigational, oral medication for the purpose of HIV PrEP
  * Willing and able to independently provide written informed consent
  * Tests HIV negative at time of screening using rapid HIV antibody test or serum antibody/antigen 4th generation HIV test
  Interventions: Drug: FTC/TAF
- Cohort 1b (Experimental): Age 18 or older at the time of signed informed consent
  * Not currently taking commercial FTC/TDF for PrEP or any other investigational, oral medication for the purpose of HIV PrEP
  * Willing and able to independently provide written informed consent
  * Tests HIV negative at time of screening using rapid HIV antibody test or serum antibody/antigen 4th generation HIV test
  Interventions: Drug: FTC/TAF
- Cohort 2 (Active Comparator): * Age 18 or older at the time of signed informed consent
  * Willing and able to independently provide written informed consent
  * Last viral load < 20 copies/mL within the last four weeks of screening
  * Must be on combination antiretroviral therapy that includes TAF/FTC for at least 6 months
  * Undetectable viral load, as defined by < 50 copies/ml, for at least 6 months
  Interventions: Drug: FTC/TAF

INTERVENTIONS:
Drug: FTC/TAF — Participants in cohorts 1a&b will be administered FTC/TAF for 1 to 7 consecutive days and then be followed clinically for 6 to 14 days. Cohort 2 will participate in a 1 time blood and urine collection.

SUMMARY:
Pre-exposure prophylaxis (PrEP) with Truvada™ (tenofovir/emtricitabine), in which an HIV-uninfected individual at high risk for contracting HIV takes antiretroviral medications (one pill daily) to maintain blood and genital drug levels sufficient to prevent HIV-1 acquisition, has been validated in several large international trials that have included men who have sex with men and transgender women, heterosexual men and women, and people who use injection drugs, as a potential HIV-1 prevention strategy. HIV prevention interventions such as this, if adequately disseminated and implemented broadly, may help to curb new HIV infections, reduce HIV-associated morbidity and mortality, and reduce health disparities in HIV rates among the most at-risk individuals. Assuring adherence to a daily dose of PrEP is critical for effective protection against HIV infection. A urine-based test to measure PrEP medication levels in the body represents a non-invasive technique to assess adherence and ultimately improve PrEP's protective ability.

TAF/FTC (Descovy™) is a new medication under study for HIV prevention to see if it is as effective as Truvada™. This study is testing whether a urine test can detect this medication in urine.

DETAILED DESCRIPTION:
Primary Objectives:

1a) To determine how long TFV is excreted in the urine in patients at steady state of TAF/FTC. Ten healthy subjects will be given seven daily doses of TAF/FTC under direct observation to ensure adherence. Morning urine and plasma samples will be collected starting the day the last is given (1 hour later) and every day thereafter for 9 days (total of 10 days of sample collection). This will allow for the assessment of the length of time TFV can be measured in the urine after last dose is taken (the "lookback" period) in the context of consistent adherence, as well as to determine how many days a patient has been off drug if a urine specimen has no detectable TFV. A correction analysis similar to that below will also be assessed in this cohort.

1b) To determine how long TFV is excreted in the urine in patients who have taken one dose of TAF/FTC. Ten healthy subjects will be given one dose of TAF/FTC under direct observation to ensure adherence. Morning urine and plasma samples will be collected starting the day the dose is given (1 hour later) and every day thereafter for 6 days (total of 7 days of sample collection). This will allow for the assessment of the length of time TFV can be measured in the urine after last dose is taken (the "lookback" period) in the context of inconsistent or intermittent (1 day only) adherence, as well as to determine how many days a patient has been off drug if a urine specimen has no detectable TFV. Investigators will also examine the correct urine TFV values for inter-subject variability by assessing which measure (specific gravity, urine creatinine, pH) will maximize the correlation between urine TFV levels and an ideal line of elimination.

Secondary Objective:

To determine the expected urine tenofovir levels in a population of HIV-positive patients on TAF-based regimens. A cross-sectional analysis of ten HIV-positive patients with undetectable viral loads on a TAF-based single tablet HIV regimen will be conducted. Morning urine and plasma samples will be collected at one time point to determine urine TFV concentration in the setting of steady state dosing in HIV patients with presumably very good adherence to medication, and compared to a historical cohort of patients on TDF-based regimens.

ELIGIBILITY:
Cohort 1(a & b) Inclusion Criteria:

* Age 18 or older at the time of signed informed consent
* Not currently taking commercial Truvada for PrEP or any other investigational, oral medication for the purpose of HIV PrEP
* Willing and able to independently provide written informed consent
* Tests HIV negative at time of screening using rapid HIV antibody test or serum antibody/antigen 4th generation HIV test

Cohort 1(a & b) Exclusion Criteria:

* Evidence of acute or chronic hepatitis B infection at the time of screening
* Other clinically significant acute or chronic medical condition, including severe infections requiring treatment such as tuberculosis, as determined by the study investigator
* Evidence of renal dysfunction (Creatinine Clearance < 30 ml/min) at the time of screening; Use Cockroft-Gault equation: GFR = (140-Age in years) x (Weight in kg) / (72 x serum creatinine)
* History of bone fractures not explained by trauma
* Grade 3 laboratory abnormality on screening tests/assessments as defined by the DAIDS grading system
* Known allergy/sensitivity to the study drug or its components
* Experiencing decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Any other clinical condition or prior therapy that, in the opinion of the Principal Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Cohort 2 Inclusion Criteria:

* Age 18 or older at the time of signed informed consent
* Willing and able to independently provide written informed consent
* Last viral load < 20 copies/mL within the last four weeks of screening
* Must be on combination antiretroviral therapy that includes TAF/FTC for at least 6 months
* Undetectable viral load, as defined by < 50 copies/ml, for at least 6 months

Cohort 2 Exclusion Criteria:

* Other clinically significant acute or chronic medical condition, including severe infections requiring treatment such as tuberculosis, as determined by the study investigator
* Evidence of renal dysfunction (Creatinine Clearance < 30 ml/min) at the time of screening; Use Cockroft-Gault equation: GFR = (140-Age in years) x (Weight in kg) / (72 x serum creatinine)
* Grade 3 laboratory abnormality on screening tests/assessments as defined by the DAIDS grading system
* Experiencing decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Any other clinical condition or prior therapy that, in the opinion of the Principal Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia FIGHT, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lalley-Chareczko L, Hiserodt E, Moorthy G, Zuppa A, Mounzer K, Koenig H. Urine Assay to Measure Tenofovir Concentrations in Patients Taking Tenofovir Alafenamide. Front Pharmacol. 2020 Mar 19;11:286. doi: 10.3389/fphar.2020.00286. eCollection 2020. PMID 32265700

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: Person living with HIV, currently prescribed an FTC/TAF based regimen, who reports recent adherence
- Cohort 1a: HIV negative adults, who are not taking FTC/TDF for PrEP; given 7 consecutive, daily doses of FTC/TAF
- Cohort 1b: HIV negative adults, who are not currently taking FTC/TDF for PrEP; administered single dose of FTC/TAF
Period: Overall Study
Arm/Group | Cohort 2 | Cohort 1a | Cohort 1b
Started | 17 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 7 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 2 | Cohort 1b | Cohort 1a | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 10 | 28
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.00 (8.88) | 30.10 (6.12) | 33.00 (9.12) | 40.03 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 8
  Male | 9 | 6 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 7
  White | 6 | 6 | 8 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Urine Samples Containing TFV in Concentrations Greater Than or Equal to 1000ng/mL From the 7-dose Cohort (1b).
Description: Cohort 1b: To determine how long TFV is excreted in the urine in patients at steady state of TAF/FTC. Ten healthy subjects will be given seven daily doses of TAF/FTC under direct observation to ensure adherence. Morning urine samples will be collected starting the day the last is given (1 hour later) and every day thereafter for 9 days (total of 10 days). Urine samples collected from all participants were analyzed via LC-MS/MS for tenofovir concentrations.
Time Frame: Daily for a maximum of 10 days
Population: 10 samples were collected each day during the sampling period (1 per participant).
Measure: Number; unit: percentage of urine samples
Units Other Than Participants: urine samples
Groups:
- Cohort 1b: HIV negative adults, who are not taking FTC/TDF for PrEP; given 7 consecutive, daily doses of FTC/TAF
Arm/Group | Cohort 1b
Number analyzed (Participants) | 10
Number analyzed (urine samples) | 100
percentage of urine samples
  Day 0 post dosing: number analyzed (urine samples) | 10
  Day 0 post dosing | 100
  Day 1 post dosing: number analyzed (urine samples) | 10
  Day 1 post dosing | 80
  Day 2 post dosing: number analyzed (urine samples) | 10
  Day 2 post dosing | 80
  Day 3 post dosing: number analyzed (urine samples) | 10
  Day 3 post dosing | 80
  Day 4 post dosing: number analyzed (urine samples) | 10
  Day 4 post dosing | 30
  Day 5 post dosing: number analyzed (urine samples) | 10
  Day 5 post dosing | 30
  Day 6 post dosing: number analyzed (urine samples) | 10
  Day 6 post dosing | 20
  Day 7 post dosing: number analyzed (urine samples) | 10
  Day 7 post dosing | 20
  Day 8 post dosing: number analyzed (urine samples) | 10
  Day 8 post dosing | 0
  Day 9 post Dosing: number analyzed (urine samples) | 10
  Day 9 post Dosing | 0

2. Primary Outcome: Percent of Urine Samples Containing TFV Levels Greater Than or Equal to 1000ng/mL in the Single Dose Cohort (1a).
Description: To determine how long TFV is excreted in the urine in patients who have taken one dose of TAF/FTC. Ten healthy subjects will be given one dose of TAF/FTC under direct observation to ensure adherence. Morning urine samples will be collected starting the day the dose is given (1 hour later) and every day thereafter for 6 days (total of 7 days of sample collection). This will allow for the assessment of the length of time TFV can be measured in the urine after last dose is taken (the "lookback" period) in the context of inconsistent or intermittent (1 day only) adherence, as well as to determine how many days a patient has been off drug if a urine specimen has no detectable TFV.
Time Frame: 7 days
Population: 10 urine samples collected on each of 7 collection days (1 per participant).
Measure: Number; unit: percentage of urine samples
Units Other Than Participants: urine samples
Groups:
- Cohort 1a: HIV negative adults, who are not currently taking FTC/TDF for PrEP; administered single dose of FTC/TAF
Arm/Group | Cohort 1a
Number analyzed (Participants) | 10
Number analyzed (urine samples) | 70
percentage of urine samples
  Day 0 post dosng: number analyzed (urine samples) | 10
  Day 0 post dosng | 60
  Day 1 post dosing: number analyzed (urine samples) | 10
  Day 1 post dosing | 60
  Day 2 post dosing: number analyzed (urine samples) | 10
  Day 2 post dosing | 30
  Day 3 post dosing: number analyzed (urine samples) | 10
  Day 3 post dosing | 20
  Day 4 post dosing: number analyzed (urine samples) | 10
  Day 4 post dosing | 0
  Day 5 post dosing: number analyzed (urine samples) | 10
  Day 5 post dosing | 0
  Day 6 post dosing: number analyzed (urine samples) | 10
  Day 6 post dosing | 10

3. Primary Outcome: Percentage of Urine Samples Containing Tenofovir at Concentrations Greater Than or Equal to 1000ng/mL (Cohort 2).
Description: To determine the expected urine tenofovir levels in a population of patients living with HIV on TAF-based regimens. A cross-sectional analysis of ten patients living with HIV with undetectable viral loads on a TAF-based single tablet HIV regimen will be conducted. Morning urine samples will be collected at one time point to determine urine TFV concentration in the setting of steady state dosing in HIV patients with presumably very good adherence to medication.
Time Frame: 1 day
Measure: Number; unit: percentage of urine samples
Units Other Than Participants: urine samples
Arm/Group | Cohort 2
Number analyzed (Participants) | 10
Number analyzed (urine samples) | 10
percentage of urine samples | 100

ADVERSE EVENTS:
Time Frame: Beginning after first dose and extending through completion of the study (Cohort 1a = 7 days; Cohort 1b = 10 days; Cohort 2 = only AEs related to blood draw collected).
Arm/Group | Cohort 2 | Cohort 1b | Cohort 1a
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2 (N=10) | Cohort 1b (N=10) | Cohort 1a (N=10)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03350672/Prot_SAP_001.pdf